CLINICAL TRIAL: NCT04279236
Title: A Prospective Multi-Center Study on the Performance of the Ponto Implant System Using Minimally Invasive Ponto Surgery (MIPS)
Brief Title: Multi-Center Study on Performance of the Ponto Implant System Using Minimally Invasive Ponto Surgery (in Adult Patients)
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC100
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-arm: In this single-arm study, the only interventions compared to routine clinical practice are the completion of two patient questionnaires (APHAB and GBI) and an additional follow-up visit after surgery.
  Interventions: Other: Abbreviated Profile Hearing Aid Benefit (APHAB); Other: Glasgow Benefit Inventory (GBI); Other: Additional follow-up visit

INTERVENTIONS:
Other: Abbreviated Profile Hearing Aid Benefit (APHAB) — An intervention in this study which is outside the routine clinical practice of the clinics is the APHAB questionnaire that will be completed by the subjects on 2 occasions.
Other: Glasgow Benefit Inventory (GBI) — An intervention in this study which is outside the routine clinical practice of the clinics is the GBI questionnaire that will be completed by the subjects on 2 occasions.
Other: Additional follow-up visit — There is an additional follow-up visit after surgery (compared to the routine clinical practice of the surgeons/clinics).

SUMMARY:
This prospective, multi-center study funded by Oticon Medical AB will be conducted at six clinical sites in North America. Patients with a hearing loss and that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study. The total number of participants included in the study will be 64.

The purpose of this study is to investigate the rate of successful BAHS use after implantation of the Ponto Implant system using the surgical technique Minimally Invasive Ponto Surgery (MIPS).

DETAILED DESCRIPTION:
This prospective, multi-centre study funded by Oticon Medical AB will be conducted at six clinical sites in North America. Patients with a hearing loss and that are already planned for treatment with a percutaneous (through the skin) bone-anchored hearing system (BAHS) will be included in the study. The total number of participants included in the study will be 64. Patients who are withdrawn from the study prior to completion will not be replaced.

The purpose of this study is to investigate the rate of successful BAHS use after implantation of the Ponto Implant system using the surgical technique Minimally Invasive Ponto Surgery (MIPS). The implant, coupled to a skin-penetrating abutment, is implanted in the bone behind the ear and is later loaded with a sound processor which transforms sound waves to sound vibrations that can be sent directly to the inner ear via the skull bone. The primary objective of this study is to investigate the proportion of implant/abutment complexes providing a reliable anchorage for a sound processor, 3 months after implantation/surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient indicated for surgical intervention with a bone anchored hearing system according to local clinic's standard guidelines.
* Normal bone quality and bone thickness above 3 mm, where no complications during surgery are expected.
* Skin thickness of 12mm or less at the implant site

Exclusion Criteria:

* Patients undergoing re-implantation
* Patients who are unable or unwilling to follow investigational procedures/requirements, e.g. to complete quality of life scales.
* Diseases or treatments known to compromise the bone quality at the implant site, e.g. radiotherapy, osteoporosis, diabetes mellitus
* Known conditions (e.g. uncontrolled diabetes) that could jeopardize skin condition and wound healing over time as judged by the investigator.
* Any other known condition that the investigator determines could interfere with compliance or study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to participating clinics who meet clinical indications for surgical intervention with a bone anchored hearing system.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Implant/abutment complex capability to provide reliable anchorage for sound processor | 3 months after implant surgery (MIPS)
  The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin over-growth and pain preventing use of the sound processor. For a positive outcome of the primary endpoint (reliable anchorage), the implant should be in place and stable. without any adverse skin reactions or skin over-growth and pain preventing usage of the sound processor.

SECONDARY OUTCOMES:
Implant/abutment complex capability to provide reliable anchorage for sound processor | 12 months after implant surgery (MIPS)
  The variables assessed to determine reliable anchorage in the study are implant survival and stability, skin reactions, skin over-growth and pain preventing use of the sound processor. For a positive outcome of the primary endpoint (reliable anchorage), the implant should be in place and stable without any adverse skin reactions or skin over-growth and pain preventing usage of the sound processor.
Implant survival | 12 months after implant surgery (MIPS)
  Implant survival will be assessed by the investigator by means of a Yes/No question: Implant/abutment complex in place [Yes/No]
Implant stability | 12 months after implant surgery (MIPS)
  Clinical assessment of implant stability by the investigator by means of a Yes/No question: Implant stable [Yes/No]
Holgers score ratings | 12 months after implant surgery (MIPS)
  Distribution of Holgers score ratings (scale 0-4) where a higher score corresponds to a poorer outcome, assigned by investigator
IPS scores | 12 months after implant surgery (MIPS)
  Distribution of IPS (Inflammation [total score 0-4], Pain [score 0-2], Skin height [score 0-2]) scores assigned by investigator. The IPS score is presented as [Ix Px Sx] with x being the individual score for each parameter. A higher score corresponds to a poorer outcome
Patient-perceived presence of pain around implant/abutment | 12 months after implant surgery (MIPS)
  Assessment of presence of patient-perceived pain by means of a Yes/No question to the subject
Patient-perceived magnitude of pain around implant/abutment | 12 months after implant surgery (MIPS)
  Assessment of magnitude of patient-perceived pain using a numerical rating scale (NRS) (range 0-10) where a higher rating corresponds to a poorer outcome
Patient-perceived presence of numbness around implant/abutment | 12 months after implant surgery (MIPS)
  Assessment of presence of patient-perceived numbness by means of a Yes/No question to the subject
Patient-perceived magnitude of numbness around implant/abutment | 12 months after implant surgery (MIPS)
  Assessment of magnitude of patient-perceived numbness using a numerical rating scale (NRS) (range 0-10) where a higher rating corresponds to a poorer outcome
Skin/soft tissue overgrowth | 12 months after implant surgery (MIPS)
  Skin overgrowth over implant/abutment complex judged by the investigator by means of a Yes/No question
Duration of surgery | At implant surgery (MIPS)
  Length of surgery measured in minutes
Wound dehiscence | 12 months after implant surgery (MIPS)
  Prevalence of wound dehiscence measured as millimeters of dehiscence
Wound healing time | 12 months after implant surgery (MIPS)
  Average healing time [days] from surgery when the wound is considered healed
Implant/abutment usage | 12 months after implant surgery (MIPS)
  Mean hours of use of a sound processor on the implant/abutment
Subjective benefit after MIPS surgery | At screening visit (visit before surgery)
  Abbreviated Profile Hearing Aid Benefit (APHAB) questionnaire score (1-99) where a global higher score corresponds to a poorer outcome
Subjective benefit after MIPS surgery | 6 months after implant surgery (MIPS)
  Abbreviated Profile Hearing Aid Benefit (APHAB) questionnaire score (1-99) where a higher global score corresponds to a poorer outcome
Subjective benefit after MIPS surgery | 3 months after implant surgery (MIPS)
  Glasgow Benefit Inventory (GBI) questionnaire score (-100 to +100) where [-100] means maximum adverse effect, [0] means no effect, and [+100] means maximum positive effect
Subjective benefit after MIPS surgery | 12 months after implant surgery (MIPS)
  Glasgow Benefit Inventory (GBI) questionnaire score (-100 to +100) where [-100] means maximum adverse effect, [0] means no effect, and [+100] means maximum positive effect

OTHER OUTCOMES:
Safety outcome | 12 months after implant surgery (MIPS)
  Occurrence and severity of both related and unrelated adverse events after MIPS surgery

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Silverstein Institute, Sarasota, Florida
  - Otolaryngology Associates, Indianapolis, Indiana
  - New York Eye and Ear Infirmary, New York, New York
  - Northwest Ear Institute, Portland, Oregon
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- The Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada
- Hospital Universitario de Donostia, San Sebastián, Gipuzkoa, Spain